Version 1.2 March 12, 2019

MONitoring of ANTI-dementia drugs by determining serum concentrations, importance of monitoring for the incidence of side effects, clinical effect and compliance ("MONANTI")

Document type: Declaration of consent

NCT number: NCT04117178

EudraCT: 2017-002707-10

Version 1.2 March 12, 2019

## Declaration of consent

Informed consent for participation in a biomedical research project

The title of the research project: MONitoring of ANTI-dementia drugs by determining serum concentrations, importance of monitoring for side effect occurrence, clinical effect and compliance ("MONANTI"). (Measurement of the blood concentration of anti-dementia drugs to improve effect and reducing side effects)

Statement from the responsible physician

I declare that the participant has received oral and written information about the research project and has had the opportunity to ask me questions. In my opinion, sufficient information has been provided for a decision to be made about participation in the trial.

| Name of the physician in charge: | |
|---|---|
| Date:Signature: | |
| Participant's statement: | |
| I have received written and oral information, and I know enough about the purp | |
| advantages and disadvantages to agree to participate. I know that participation is I can always withdraw my consent without losing my current or future rights to | • |
| to participate in the research project and I have received a copy of this consent | |
| the written information about the project for my own use. | |
| I want to be information about my health that may become evident during the s | tudy: Yes □ No □ |
| I wish to receive information about the results of the current examination: | |
| Yes □ No □ | |
| Name of the participant: | (capital letters) |
| Date:Signature: | |